CLINICAL TRIAL: NCT05753059
Title: Mechanisms of Diuretic Resistance in Heart Failure, Aim 2
Acronym: MsDR 2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey Testani, Associate Professor of Medicine, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000034315; 1R01DK130997-01 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Amiloride; Bendroflumethiazide

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled, double-blind, double-dummy, crossover design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo/ Placebo (Placebo Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Interventions: Drug: Placebo
- Placebo/ Amiloride (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Interventions: Drug: Placebo; Drug: Amiloride
- Placebo/ Bendroflumethiazide (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Interventions: Drug: Placebo; Drug: Bendroflumethiazide
- Bendroflumethiazide/ Amiloride (Active Comparator): This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Interventions: Drug: Amiloride; Drug: Bendroflumethiazide

INTERVENTIONS:
Drug: Placebo — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, added to bumetanide on Days 0, 7, 14 and 21
  Arms: Placebo/ Amiloride; Placebo/ Bendroflumethiazide; Placebo/ Placebo
Drug: Amiloride — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations of amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Arms: Bendroflumethiazide/ Amiloride; Placebo/ Amiloride
Drug: Bendroflumethiazide — This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations of bendroflumethiazide/placebo and bendroflumethiazide/amiloride added to bumetanide on Days 0, 7, 14 and 21
  Arms: Bendroflumethiazide/ Amiloride; Placebo/ Bendroflumethiazide

SUMMARY:
Randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide.

DETAILED DESCRIPTION:
This study will employ a randomized placebo-controlled, double-blind, double-dummy, crossover design testing combinations placebo/placebo, bendroflumethiazide/placebo, amiloride/placebo, and bendroflumethiazide/amiloride added to bumetanide.

Patients will be co-enrolled in this study and an ancillary study for administration of Bendroflumethiazide. Administration of bendroflumethiazide will take place under an ancillary protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of HF
2. No plan for titration/change of heart failure medical or device therapies during the study period.
3. Absence of non-elective hospitalizations in the previous 2 weeks
4. At optimal volume status by symptoms, exam, and dry weight.
5. Serum potassium ≤ 5.0 mmol/L
6. Serum sodium ≥ 130 mEq/L
7. Age > 18 years
8. Hemoglobin ≥8 g/dL
9. Objective evidence of diuretic resistance to a 10mg bumetanide challenge, defined as:

   1. FENa <10% and total sodium output <150mmol and
   2. At least one of the following criteria:

1. Chronic home furosemide dose > or equal to 80mg furosemide equivalents daily 2. eGFR < 60ml/min 3. Serum chloride <100mmol/L 4. FENa <5% and total sodium output <75mmol on the 2 hour screening

Exclusion Criteria:

1. GFR <20 ml/min/1.73m2 using the CKD-EPI equation or use of renal replacement therapies
2. Use of any non-loop type diuretic in the last 7 days or 5 half lives, with the exclusion of low dose aldosterone antagonist (e.g., spironolactone or eplerenone ≤50 mg). Examples of non-loop diuretics include but may not be limited to acetazolamide (oral or IV, not ophthalmic), metolazone, HCTZ, chlorthalidone, chlorothiazide, indapamide, triamterene, amiloride, finerenone, spironolactone dose > 50mg day, eplerenone > 50mg/day,
3. History of flash pulmonary edema requiring hospitalization and treatment with biphasic positive airway pressure or mechanical ventilation or a "brittle" volume sensitive HF phenotype such as an infiltrative or restrictive cardiomyopathy (i.e. amyloid cardiomyopathy, etc).
4. Hemoglobin < 8 g/dL or symptomatic anemia
5. Pregnant or breastfeeding
6. Inability to give written informed consent or comply with study protocol or follow-up visits
7. Chronic urinary retention limiting ability to perform timed urine collection procedures
8. On Lithium therapy
9. On pimozide or thioridazine
10. Diagnosis of liver failure
11. Contraindications or allergy to sulfonamides
12. Any contraindication to thiazide diuretic or allergy to thiazide or bendroflumethiazide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in peak FENa from bumetanide monotherapy to bumetanide plus combination therapy | 21 days
  Change in peak FENa from bumetanide monotherapy to bumetanide plus combination therapy
Change in distal sodium reabsorption | 21 days
  Change in distal sodium reabsorption (FELi minus FENa) from bumetanide monotherapy to bumetanide plus combination therapy
Correlation between distal sodium reabsorption and uEV pendrin/CD9 | 21 days
  Correlation between distal sodium reabsorption (FELi minus FENa) and uEV pendrin/CD9

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No